CLINICAL TRIAL: NCT07205614
Title: The Good Pain Consultation in Endometriosis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 813570; 818856 (Other: Regional Committes for Medical and Health Research Ethics South-East Norway)
Record Dates: First submitted 2025-09-17; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Pelvic Pain Syndrome; Endometriosis; Dysmenorrhea; Adenomyosis; Period Pain; Menstrual Pain
Keywords: pain education; biopsychosocial; randomised controlled trial
MeSH Terms: conditions — Endometriosis; Dysmenorrhea; Adenomyosis

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinded outcome assessment and data analysis. Manuscript first draft will be written blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): pain consultation, biopsychosocial pain education + usual care
  Interventions: Other: pain consultation, biopsychosocial pain education + usual care
- control group (Other): usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: pain consultation, biopsychosocial pain education + usual care — Participants will receive a link to a digital pain education program. The program will include standard information about endometriosis, but will also introduce a biopsychosocial understanding of pain including influence of psychological factors such as excessive worry, stress, sleep disturbance and emotional distress. Self-management strategies including physical activity, relaxation and breathing techniques, cognitive techniques, psychosocial support and appropriate use of pain medication and supplemental treatment (e.g. physical therapy, TENS, heat), will be introduced.
  Participants will then attend a single "good pain consultation", a patient-centered consultation with a clinician associated with the project, in which content from the educational package will be reinforced. The consultation will provide the opportunity to address the biopsychosocial factors including anxiety, previous trauma, emotional distress etc. Shared decision-making regarding preferred self-management strat
  Arms: intervention group
Other: Usual Care — Usual follow up at the department of gynecology
  Arms: control group

SUMMARY:
This PhD project investigates the effect of "the good pain consultation" and early integration of biopsychosocial pain education with current standard management of endometriosis. Our goal is to facilitate self-management of pain and improve health-related quality of life (HRQOL) using limited resources.

Our research question is: Does a good pain consultation improve pain self-efficacy and HRQOL, compared to usual care at 3 months and 1 year.?

Researchers will compare a good pain consultation to a control group that will receive usual care.

Participants will:

Attend a consultation and biopsychososial pain education plus usual care or usual care alone.

They will answer questions in an internet-based questionnaires three times point during the study.

ELIGIBILITY:
Inclusion Criteria:

* biological women

Exclusion Criteria:

* not speaking norwegian

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
The Pain Self-Efficacy Questionaire | The participants will report the outcome measures at baseline, after 3 and after 12 months.
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10 item self-report questionnaire which assesses confidence people with ongoing pain have in performing activities despite pain. Self-efficacy regarding household chores, socializing, work and coping without medication are assessed. Each item is scored on a 6-point scale, for a total raw score of 0-10 where high scores indicate greater levels of confidence in dealing with pain. The PSEQ is translated to Norwegian and used in previous Norwegian studies.

SECONDARY OUTCOMES:
The Short Form-12/Rand 12 Health Survey | The participants will report the outcome measures at baseline, after 3 and after 12 months.
  SF-12 is a tool for assessing HRQOL, encompassing eight health domains: physical functioning, role limitations due to physical and emotional problems, bodily pain, general health, vitality, social functioning, and mental health. These domains form two summary measures: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).
A single question about Quality of Life | The participants will report the outcome measures at baseline, after 3 and after 12 months.
  They will be asked: "All in all, how satisfied are you with your life right now?" we are using a scale from 0 to 10, where 0 means not at all satisfied and 10 means very satisfied.
Pain catastrophizing scale (PCS) | The participants will report the outcome measures at baseline, after 3 and after 12 months.
  PCS measures pain catastrophizing and "exaggerated negative orientation toward pain stimuli and pain experience". The scale consists of 13 items and includes subscale scores for rumination, magnification and helplessness.
The Hopkins Symptom Checklist (HSCL-10). | The participants will report the outcome measures at baseline, after 3 and after 12 months.
  The Hopkins Symptom Checklist (HSCL-10) is assessing emotional distress. The HSCL-10 consists of 10 questions assessing symptoms of anxiety and depression (range 1 to 4, most symptoms). Scores ≥1.75 are indicative of increased emotional distress.
Numeric rating scales (NRS) | The participants will report the outcome measures at baseline, after 3 and after 12 months.
  Numeric rating scales (NRS) rating from 0 to 10 measuring pain intensity. 0 means no pain and 10 means worst possible pain. Three NRS measures will be done registering worst pain intensity and bothersomeness of pain, during the past month
The Decreased Sexual Desire Screener (DSDS) | The participants will report the outcome measures at baseline, after 3 and after 12 months.
  (DSDS) is a simple, validated diagnostic tool to help to identify and discuss hypoactive sexual dysfunction among women.
The Brief Illness Perception Questionnaire (Brief IPQ) | The participants will report the outcome measures at baseline, after 3 and after 12 months.
  Brief IPQ is used to assess the cognitive and emotional perception of their illness and consists of nine questions. Answers are scored on a Likert scale from 0-10 scale in the first eight question and the latter question has an open-ended respons. Higher scores indicate more threatening/negative views of their pelvic pain.
2016 Fibromyalgia diagnostic criteria | The participants will report the outcome measures at baseline, after 3 and after 12 months.
  The 2016 Fibromyalgia diagnostic criteria are used to identify fibromyalgia based on symptom severity and pain distribution. The criteria include two main components:
  * Widespread Pain Index (WPI), which Assess pain in 19 body regions over the past week with a Score range: 0-19 (1 point per painful area)
  * Symptom Severity Scale (SSS) measures severity (0-3) of fatigue, unrefreshing sleep, and cognitive symptoms with a score range: 0-12
  Diagnosis is met if: WPI ≥ 7 and SSS ≥ 5, or WPI 4-6 and SSS ≥ 9 and symptoms have been present at a similar level for at least 3 months, with generalized pain in at least 4 of 5 body regions
Other questions | The participants will report the outcome measures at baseline and after 12 months.
  We will ask questions about sociodemographic factors, symptoms related to the condition, and how one lives with the condition. Additionally, medical record information regarding the current condition and comorbidity
intention to reconsult and use of healthcare services | The participants will report the outcome measures at baseline and after 12 months
  Intention to re-consult, use of health care services and use of medication will be elicited. The partisipant will report this in questionaires, and data will also be collected from national registers.

CONTACTS AND LOCATIONS:
Locations (1):
- Sorlandet Sykehus HF, Kristiansand, Agder, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-09-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT07205614/Prot_SAP_ICF_000.pdf